CLINICAL TRIAL: NCT00821470
Title: Treatment of Osteonecrosis of the Femoral Head With Implantation of Autologous Bone Marrow Cells, a Pilot Study
Brief Title: Treatment of Osteonecrosis of the Femoral Head by Bone Marrow Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Responsible Party: Valerie Gangji, Erasme Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ref. 98/20
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Necrosis
Keywords: osteonecrosis; bone marrow; core decompression; femoral head
MeSH Terms: conditions — Necrosis; Osteonecrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bone marrow graft group (Experimental): core decompression + bone marrow implantation into the necrotic lesion
  Interventions: Procedure: core decompression; Procedure: Bone marrow implantation into the necrotic lesion
- control (Active Comparator): core decompression
  Interventions: Procedure: core decompression

INTERVENTIONS:
Procedure: core decompression — core decompression procedure only
Procedure: Bone marrow implantation into the necrotic lesion
  Arms: bone marrow graft group

SUMMARY:
Aseptic non traumatic osteonecrosis (ON) is a painful disorder of the hip which often leads, in its final stage, to femoral head collapse and subsequent total hip replacement. Core decompression of the hip is the most widespread procedure used to treat early stage ON of the femoral head. Notwithstanding the fact that this procedure has been employed for more than three decades (2), its efficacy remains controversial (3;4). Recently, one suggested that ON might be a disease of bone cells and/or of mesenchymal cells. The levels of activity and the number of mesenchymal stem cells in both the hematopoietic and in the stromal compartments of the bone marrow have been shown to be depressed in patients with ON of the femoral head (9). The investigators have showed previously that the capacity of osteoblastic cells to replicate was decreased in the proximal femur of patients with ON of the femoral head (10). This finding raised the possibility that bone marrow containing stromal cells which have many of the characteristics of stem cell for mesenchymal tissues including bone could be implanted into the necrotic lesion of the femoral head.

ELIGIBILITY:
Inclusion Criteria:

* ARCO stage 1 or 2 osteonecrosis of the femoral head

Exclusion Criteria:

* The investigators excluded patients with evidence of a malignant disorder during the past five years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 1999-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
WOMAC Score | 60 months

SECONDARY OUTCOMES:
Disease progression defined as progression to a fractural stage of osteonecrosis | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: valerie gangji, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels, Belgium